CLINICAL TRIAL: NCT07253740
Title: Comparison of Interscalene and Infraspinatus-Teres Minor Blocks on Postoperative Opioid Consumption and Pain Scores in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Interscalene Versus Infraspinatus-Teres Minor Blocks for Arthroscopic Shoulder Surgery
Acronym: ITM-ISB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator Ali Ahıskalıoğlu, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATAUNISHOULDER
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: Postoperative Pain; Analgesia; Regional Anesthesia; Interscalene Brachial Plexus Block; Infraspinatus-Teres Minor Block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist performing the blocks is aware of the group allocation; all other staff and outcome assessors are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Brachial Plexus Block (ISB) (Experimental): Patients will receive ISB under ultrasound guidance prior to arthroscopic shoulder surgery using 15 ml 0.25% bupivacaine.
  Interventions: Procedure: Interscalene Brachial Plexus Block (ISB)
- Infraspinatus-Teres Minor Block (ITM) (Experimental): Patients will receive TM block under ultrasound guidance using 25 ml 0.25% bupivacaine between infraspinatus and teres minor muscles.
  Interventions: Procedure: Infraspinatus-Teres Minor Block (ITM)

INTERVENTIONS:
Procedure: Interscalene Brachial Plexus Block (ISB) — Patients receive ultrasound-guided ISB before arthroscopic shoulder surgery. After sedation with IV midazolam, 15 ml of 0.25% bupivacaine is injected using a 22 Gauge 50 mm needle with posterior in-plane approach, targeting C5-C6 roots.
  Other Names: Interscalene Nerve Block
  Arms: Interscalene Brachial Plexus Block (ISB)
Procedure: Infraspinatus-Teres Minor Block (ITM) — Patients receive ultrasound-guided ITM interfascial block in sitting position before surgery. Using a 22 Gauge 10 mm needle, 25 ml of 0.25% bupivacaine is injected between infraspinatus and teres minor muscles via out-of-plane or in-plane hydrodissection.
  Arms: Infraspinatus-Teres Minor Block (ITM)

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of interscalene (ISB) and infraspinatus-teres minor (ITM) blocks for postoperative analgesia in patients undergoing elective arthroscopic shoulder surgery. The primary outcome is total 24-hour opioid consumption. Secondary outcomes include pain scores, hemidiaphragmatic paresis incidence and severity, duration of analgesia, and changes in lung function. Participants are randomized into ISB or ITM groups; blocks are performed under ultrasound guidance. Postoperative pain is managed with patient controlled analgesia(PCA).

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized clinical trial designed to compare the efficacy of Interscalene Brachial Plexus Block (ISB) and Infraspinatus-Teres Minor (ITM) interfascial block in patients undergoing elective unilateral arthroscopic shoulder surgery. The primary objective is to compare total 24-hour postoperative opioid consumption. Secondary objectives include the and pain scores, incidence and severity of hemidiaphragmatic paresis, duration of analgesia (from block completion to initiation of IV PCA), and postoperative pulmonary function changes.

This study aims to determine whether the ITM block provides comparable perioperative analgesia to the ISB block while potentially reducing hemidiaphragmatic paresis and pulmonary compromise.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists I-III
* Scheduled for elective unilateral arthroscopic shoulder surgery
* Provide written informed consent

Exclusion Criteria:

* Refusal to participate
* Allergy to study drugs
* Severe cardiac, renal, or hepatic disease
* Neurological deficit or neuropathy
* Anticoagulant therapy
* Pre-existing respiratory dysfunction
* Chronic shoulder pain or planned open surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Total 24-Hour Postoperative Opioid Consumption | 0-24 hours postoperatively
  Total intravenous opioid consumption recorded for each patient during the first 24 hours after arthroscopic shoulder surgery, including any rescue analgesia administered.

SECONDARY OUTCOMES:
Incidence and Severity of Hemidiaphragmatic Paresis | Pre-block and 30 minutes post-block
  Ipsilateral hemidiaphragmatic function evaluated by M-mode ultrasonography before block and 30 minutes after block completion. Paresis classified as none (<25% reduction), partial (25-75% reduction), or complete (>75% reduction or paradoxical movement).
Duration of Analgesia | 0-24 hours post-block
  Time interval from block completion to initiation of IV PCA fentanyl in each patient.
Pulmonary Function Changes (FEV1) | Pre-block and 30 minutes post-block
  Pulmonary function measured with bedside spirometry pre-block and 30 minutes post-block. Forced expiratory volume in 1 second (FEV1) recorded; each measurement performed three times and mean value used.
Pulmonary Function Changes (FVC) | Pre-block and 30 minutes post-block
  Pulmonary function measured with bedside spirometry pre-block and 30 minutes post-block. Forced vital capacity (FVC) recorded; each measurement performed three times and mean value used.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahıskalıoğlu, Professor, Principal Investigator — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy concerns and institutional regulations. Data will be securely stored and used solely for the purposes of this study and related scientific publications.

REFERENCES:
- [Background] Renes SH, Rettig HC, Gielen MJ, Wilder-Smith OH, van Geffen GJ. Ultrasound-guided low-dose interscalene brachial plexus block reduces the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):498-502. doi: 10.1097/AAP.0b013e3181b49256. PMID 19920426
- [Background] Kim SH, Yeo IS, Jang J, Jung HE, Chun YM, Yang HM. Infraspinatus-teres minor (ITM) interfascial block: a novel approach for combined suprascapular and axillary nerve block. Reg Anesth Pain Med. 2024 Jan 11;49(1):67-72. doi: 10.1136/rapm-2023-104738. PMID 37491150
- [Background] Kang R, Jeong JS, Chin KJ, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Ko JS. Superior Trunk Block Provides Noninferior Analgesia Compared with Interscalene Brachial Plexus Block in Arthroscopic Shoulder Surgery. Anesthesiology. 2019 Dec;131(6):1316-1326. doi: 10.1097/ALN.0000000000002919. PMID 31490292
- [Background] Teske LG, Pill SG, Lutz A, Thigpen CA, Shanley E, Adams KJ, Bohon H, Graham GD, Marston G, Walker KB, Kissenberth MJ. Single shot interscalene regional anesthesia provides noninferior analgesia and decreased complications compared with an indwelling catheter for arthroscopic and reconstructive shoulder surgery. J Shoulder Elbow Surg. 2022 Jun;31(6S):S152-S157. doi: 10.1016/j.jse.2022.02.004. Epub 2022 Mar 15. PMID 35301140
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Luan H, Hao C, Li H, Zhang X, Zhao Z, Zhu P. Effect of interscalene brachial plexus block with dexmedetomidine and ropivacaine on postoperative analgesia in patients undergoing arthroscopic shoulder surgery: a randomized controlled clinical trial. Trials. 2023 Jun 12;24(1):392. doi: 10.1186/s13063-023-07292-2. PMID 37308994
- [Background] Ahiskalioglu A, Karapinar YE, Dagci Y, Yayik AM, Ciftci B, Tulgar S. An alternative sonographic approach to infraspinatus-teres minor interfascial plane block: make it easy. Minerva Anestesiol. 2025 Apr;91(4):359-361. doi: 10.23736/S0375-9393.24.18697-X. Epub 2025 Feb 6. No abstract available. PMID 39912574